CLINICAL TRIAL: NCT03440398
Title: Robotic Nipple-Sparing Mastectomy And Immediate Robotic Breast Reconstruction Vs Conventional Open Technique: A Prospective Randomized Trial Evaluating Patients Satisfaction
Brief Title: Robotic Nipple-Sparing Mastectomy Vs Conventional Open Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R 530/16- IEO 562
Record Dates: First submitted 2017-03-11; First posted 2018-02-22 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: Robotic Mastectomy; Nipple Sparing Mastectomy; Conservative mastectomy; Breast reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open NSM (Active Comparator): Conventional Nipple Sparing Mastectomy
  Interventions: Procedure: Open NSM
- Robotic NSM (Experimental): Robotic Nipple-Sparing Mastectomy
  Interventions: Procedure: Robotic NSM

INTERVENTIONS:
Procedure: Robotic NSM — Surgical technique conducted using robot to perform nipple sparing mastectomy and breast reconstruction
  Arms: Robotic NSM
Procedure: Open NSM — Open nipple-sparing mastectomy and immediate breast reconstruction with implant
  Arms: Open NSM

SUMMARY:
This trial is designed to compare robotic nipple-sparing mastectomy and immediate robotic breast reconstruction with conventional open technique. It is a prospective randomized trial evaluating patients satisfaction

DETAILED DESCRIPTION:
High proportion of patients with newly diagnosed early-stage breast cancer in Europe and US undergo to mastectomy. The absolute numbers of mastectomy rates in US is still today around 38% and represent one of the most performed operation for cancer reasons. Despite the lack of a natural cavity needed for endoscopic viewing, applications of robotic surgery have recently emerged for superficial organs such as in the fields of thyroidectomy, oropharyngeal surgery, plastic and reconstructive surgery. However, it has never been applied in breast cancer except for a feasibility and safety study conducted at European Institute of Oncology.

The technique was firstly published by Toesca et al. considering the first 3 cases. The same research as continued on breast cancer evaluating feasibility, reproducibility and safety studying 26 consecutive procedures of robotic nipple sparing mastectomy and immediate robotic breast reconstruction (article under peer to peer review at European Journal of Surgical Oncology, EJSO). In these initial cases of robotic nipple sparing mastectomy and immediate breast reconstruction authors found two main advantages such as the robotic optical vision and the minimal invasiveness. The two main limitations noticed in this initial experience were the duration of operating time and the additional costs related to the operation. The limitations of the applicability of robotic surgery to the breast, such as operating time and costs, might be offset by the advantages they observed such as better vision and minimally invasive approach with an anatomically more respectful mastectomy.

This project is a superiority trial comparing robotic nipple sparing mastectomy and immediate breast robotic reconstruction with conventional open technique.

The primary end-point is to evaluate patient satisfaction. Second end-point is to compare post-operative outcome considering complications, post-operative pain, reduction of the average length of stay of patients, long term oncological outcome of the two different surgical techniques.

Patients will be randomized into two treatment arms:

A. Open nipple-sparing mastectomy and immediate breast reconstruction with implant (Open NSM) B. Robotic nipple-sparing mastectomy and immediate robotic breast reconstruction with implant (Robotic NSM) Both arms will undergo to the same pre-surgical staging, intra-operative axillary surgical staging, post-operative multidisciplinary evaluation and adjuvant treatments according to international and internal protocols.

ELIGIBILITY:
Inclusion Criteria:

* Invasive breast cancer, Ductal Carcinoma In Situ, Breast Related Cancer Antigens mutation carriers.
* Any age
* Candidates to nipple-sparing mastectomy and immediate breast reconstruction
* Negative preoperative assessment of nipple-areola complex
* Absence of skin involvement
* Low probability to have positivity of nipple-areola complex tissue intra-operative frozen section
* Breast volume ≤ Bra IV; from cup A to D
* No hard smoking (hard smoking defined as >20 cigarettes/day)
* Low and intermediate risk for anesthesia (ASA Scale)
* Written informed consent must be signed and dated by the patient and the investigator prior to inclusion
* Patients must be accessible for follow-up

Exclusion criteria:

* Previous thoracic radiation therapy for any reason
* Inflammatory Breast Cancer
* Skin involvement
* Pre-operative diagnosis (radiological or cytological) of nipple-areola complex disease
* Pregnancy
* Patients with psychiatric, addictive, or any disorder, which compromises ability to give informed consent for participation in this study
* Uncompensated Diabetes Mellitus
* Hard smokers (hard smoking defined as >20 cigarettes/day)
* High risk for anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2023-12-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | 1 year
  The BREAST-Q survey is used to detect differences in patient satisfaction among the groups

SECONDARY OUTCOMES:
Average length of stay of patients | 1 month
  Reduction of the average length of stay of patients of the two different surgical techniques.
Post operative complications | 1 month
  Compare post operative complications (pain, skin or nipple-areola injury or necrosis or infection, hematoma, seroma)
Cumulative incidence of local recurrence | 5 years
  Cumulative incidence of local recurrence
Cumulative incidence of axillary recurrences | 5 years
  Cumulative incidence of axillary recurrences
Cumulative incidence of distant recurrences | 5 years
  Cumulative incidence of distant recurrences
Disease free survival | 5 years
  Disease free survival
Overall survival | 5 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Toesca, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Toesca A, Peradze N, Manconi A, Galimberti V, Intra M, Colleoni M, Bonanni B, Curigliano G, Rietjens M, Viale G, Sacchini V, Veronesi P. Robotic nipple-sparing mastectomy for the treatment of breast cancer: Feasibility and safety study. Breast. 2017 Feb;31:51-56. doi: 10.1016/j.breast.2016.10.009. Epub 2016 Nov 2. PMID 27810700
- [Result] Toesca A, Peradze N, Manconi A, Nevola Teixeira LF. Reply to the letter to the editor "Robotic-assisted Nipple Sparing Mastectomy: A feasibility study on cadaveric models" by Sarfati B. et al. J Plast Reconstr Aesthet Surg. 2017 Apr;70(4):558-560. doi: 10.1016/j.bjps.2016.12.022. Epub 2017 Jan 23. No abstract available. PMID 28153430
- [Result] Toesca A, Peradze N, Galimberti V, Manconi A, Intra M, Gentilini O, Sances D, Negri D, Veronesi G, Rietjens M, Zurrida S, Luini A, Veronesi U, Veronesi P. Robotic Nipple-sparing Mastectomy and Immediate Breast Reconstruction With Implant: First Report of Surgical Technique. Ann Surg. 2017 Aug;266(2):e28-e30. doi: 10.1097/SLA.0000000000001397. No abstract available. PMID 28692558
- [Derived] Toesca A, Sangalli C, Maisonneuve P, Massari G, Girardi A, Baker JL, Lissidini G, Invento A, Farante G, Corso G, Rietjens M, Peradze N, Gottardi A, Magnoni F, Bottiglieri L, Lazzeroni M, Montagna E, Labo P, Orecchia R, Galimberti V, Intra M, Sacchini V, Veronesi P. A Randomized Trial of Robotic Mastectomy Versus Open Surgery in Women With Breast Cancer or BrCA Mutation. Ann Surg. 2022 Jul 1;276(1):11-19. doi: 10.1097/SLA.0000000000004969. Epub 2021 Jun 9. PMID 34597010
- See also: Interview to Dr Toesca — https://www.youtube.com/watch?v=VRWXcuUBZNU&feature=youtu.be
- See also: Article on "La Repubblica" — http://la.repubblica.it/saluteseno/news/un-robot-per-curare-il-seno/5654/?refresh_ce